CLINICAL TRIAL: NCT06177379
Title: Magnetic Resonance Neurography Analysis of Healthy Human Thoracic Dorsal Root Ganglion
Status: Completed | Type: Observational
Sponsor: Huazhong University of Science and Technology (Other)
Responsible Party: Principal Investigator, Xianwei Zhang，MD, Clinical Professor, Huazhong University of Science and Technology
Other Study IDs: dorsal root ganglion
Record Dates: First submitted 2023-12-11; First posted 2023-12-20 (Actual); Last update posted 2023-12-20 (Actual); Status verified 2023-12

CONDITIONS: Dorsal Root Ganglion
Keywords: dorsal root ganglion,; Magnetic resonance neurography; volume; neuropathic pain
MeSH Terms: conditions — Neuralgia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: healthy volunteer — Volunteers age between 50 and 75 years

SUMMARY:
Here, this study aimed to conduct magnetic resonance neurography (MRN) of the thoracic DRGs in a cohort of healthy individuals. The acquired images will be thoroughly analyzed utilizing 3D-slicer software. We expect to furnish crucial baseline anatomical data of thoracic DRGs in healthy subjects, provide an anatomical basis for clinical investigation and therapeutic interventions.

DETAILED DESCRIPTION:
Chronic neuropathic pain remains a world's public health challenges, affecting hundreds of millions of people worldwide. It is estimated that 11.2% of general-practice patients suffer from neuropathic pain, and many continue to suffer from intractable pain and/or undesirable side effects. Neuropathic pain refers to the entire somatosensory system, encompassing both central and peripheral neuropathic pain. In recent years, although significant advancements have been achieved in the mechanism and management of neuropathic pain, and numerous pharmaceutical agents and therapeutic approaches have been utilized for its treatment, the outcomes still to be less than optimal. Moreover, the adverse side effects associated with certain first- and second-line medications, such as antidepressants and anticonvulsants, as well as the potential for opioid addiction, significantly impact patients' adherence to treatment. Hence, there remains a need for continued investigation into effective strategies for the management of neuropathic pain.

Therapies focused on the dorsal root ganglion (DRG) have emerged as a significant intervention in the clinical practice of pain physicians for the management of chronic pain, given its integral and important role in the signals transmission from the peripheral nervous system to the central nervous system. Accurate positioning holds paramount importance during the treatment process, necessitating clinicians to possess a comprehensive understanding of the morphology, distribution, and interconnections of the dorsal root ganglia across various segments. Currently, there exists a limited number of in vivo investigations concerning the dorsal root ganglion (DRG), with a predominant emphasis on the lumbar segment, which have mostly used invasive neuroradiography. The investigation on thoracic DRG remains largely unexplored. However, herpes zoster, the most prevalent form of neuropathic pain, manifests most frequently in the thoracic segment. Furthermore, the studies of herpes zoster reveal that DRG plays a significant role in the progression of the disease and the transmission of pain signals. Hence, a comprehensive comprehension of the anatomy and variability of thoracic DRGs assumes significance not only in accurately comprehending the pathological anatomy of neuropathic pain in the thoracic region, but also in providing guidance for interventional and individualized treatment targeting the DRGs.

ELIGIBILITY:
Inclusion Criteria:

1. age between 40 and 75 years;
2. height between 145cm to 180cm;
3. BMI between 18.5 to 30.

Exclusion Criteria:

1. scoliosis;
2. history of thoracic surgery and pain;
3. history of spinal trauma and surgery;
4. failure or inability to complete magnetic resonance neurography (MRN) scans.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: healthy volunteers aged between 50 and 75 years, height between 145cm to 180cm, and BMI between 18.5 to 30.
Sampling Method: Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-08-31 (Actual); Study Completion 2023-12-10 (Actual)

PRIMARY OUTCOMES:
the average DRG volume of healthy volunteers | 202301-202312
  the average DRG volume in each thoracic segment of healthy volunteers

SECONDARY OUTCOMES:
width/length ratio of DRGs | 202301-202312
  width/length ratio of DRGs in the slice of largest volume

CONTACTS AND LOCATIONS:
Overall Officials: Xianwei Zhang, Doctor, Principal Investigator — Huazhong University of Science and Technology
Locations (1):
- Tongji Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Attal N, Bouhassira D. Advances in the treatment of neuropathic pain. Curr Opin Neurol. 2021 Oct 1;34(5):631-637. doi: 10.1097/WCO.0000000000000980. PMID 34310363
- [Background] Berger AA, Liu Y, Possoit H, Rogers AC, Moore W, Gress K, Cornett EM, Kaye AD, Imani F, Sadegi K, Varrassi G, Viswanath O, Urits I. Dorsal Root Ganglion (DRG) and Chronic Pain. Anesth Pain Med. 2021 Mar 28;11(2):e113020. doi: 10.5812/aapm.113020. eCollection 2021 Apr. PMID 34336621
- [Background] Malik KM, Imani F, Beckerly R, Chovatiya R. Risk of Opioid Use Disorder from Exposure to Opioids in the Perioperative Period: A Systematic Review. Anesth Pain Med. 2020 Feb 19;10(1):e101339. doi: 10.5812/aapm.101339. eCollection 2020 Feb. PMID 32337175
- [Background] Attal N, Bouhassira D, Baron R. Diagnosis and assessment of neuropathic pain through questionnaires. Lancet Neurol. 2018 May;17(5):456-466. doi: 10.1016/S1474-4422(18)30071-1. Epub 2018 Mar 26. PMID 29598922
- [Background] Liem L, van Dongen E, Huygen FJ, Staats P, Kramer J. The Dorsal Root Ganglion as a Therapeutic Target for Chronic Pain. Reg Anesth Pain Med. 2016 Jul-Aug;41(4):511-9. doi: 10.1097/AAP.0000000000000408. PMID 27224659
- [Background] Bannister K, Sachau J, Baron R, Dickenson AH. Neuropathic Pain: Mechanism-Based Therapeutics. Annu Rev Pharmacol Toxicol. 2020 Jan 6;60:257-274. doi: 10.1146/annurev-pharmtox-010818-021524. PMID 31914896